CLINICAL TRIAL: NCT05536336
Title: A Randomized, Double-Blinded, Crossover and Multi-center Clinical Study to Evaluate the Performance of Synthetic Polyurethane Male Condom Compared to Standard Latex Condom During Vaginal Intercourse
Brief Title: Clinical Study to Evaluate the Performance of Synthetic Polyurethane Male Condoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor has opted to discontinue the study due to site non-compliance.
Sponsor: Okamoto Industries, Inc. (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-06
Record Dates: First submitted 2022-01-31; First posted 2022-09-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Performance of Synthetic Polyurethane Male Condom
Keywords: condom
MeSH Terms: interventions — Condoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Okamoto Lubricated Synthetic Polyurethane Male Condom (Experimental): The test device name is Okamoto 001 Lubricated Polyurethane Male Condom. The condom is made in Japan and conforms to ASTM D6324-11 (2017) Standard Test Methods for Male Condoms Made from Polyurethane.
  Interventions: Device: Condom
- Latex condom (Active Comparator): Commercially available latex lubricated condom.
  Interventions: Device: Condom

INTERVENTIONS:
Device: Condom — Contraception

SUMMARY:
This study is a randomized, double-blinded, crossover and multi-center study to evaluate the clinical breakage and slippage of a new synthetic polyurethane male condom compared to a commercially available standard latex condom.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, crossover and multi-center study to evaluate the clinical breakage and slippage of a new synthetic polyurethane male condom compared to a commercially available standard latex condom.

The duration of participation for each couple is approximately 6 weeks. Study subjects are given a set of one condom type to use for up to three consecutive weeks to complete each evaluation and then return for a set of the other condom type for another period of up to three weeks of evaluation.

The primary objective of this study is to determine whether the total clinical failure rate of a new test condom is comparable with the total clinical failure rate of a legally marketed latex condom when used during vaginal intercourse.

The secondary objective of this study is to evaluate the clinical slippage and breakage of the polyurethane and latex condoms, as well as user acceptance about using the devices and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet ALL of the following criteria for randomization into the study:

1. mutually monogamous, current relationship ≥ 3 months;
2. 18 years to 65 years of age;
3. sexually active, sufficient to meet protocol requirements; agree to have penile-vaginal intercourse with frequency sufficient to meet protocol requirements;
4. agree to use only study condoms during time of participation;
5. agree not to use drugs, ointments or non-study devices that can affect sexual performance or might affect the condom's physical property;
6. able to understand instructions for correct use of condoms;
7. no known sexually transmitted infections including HIV/AIDS;
8. agree to use only lubricant(s) provided by the study;
9. agree to return any unopened condoms and lubricants;
10. agree not to wear any genital piercing jewelry while using study condoms;

l) willing to use the study products for minimum of 10 acts of vaginal intercourse within 6 weeks of study entry; l) willing and capable of following requirements of protocol, including willingness to respond to questions about reproductive and contraceptive history and use of condoms during interviews; m) agree to use and has internet/web access in order to complete the Diaries and Surveys using iMedNet's ePRO module; n) available for follow-up and reachable by telephone.

Exclusion Criteria:

Subjects will be excluded in ANY of the following exclusion criteria apply at the time of entry or at the time during the study. If either partner is (or becomes) aware that:

1. he/she is allergic or sensitive to natural rubber latex or polyurethane,
2. female partner is pregnant or desires to become so while participating in study,
3. subject knowingly has a sexually transmitted infection,
4. commercial sex workers,
5. itinerant persons who cannot be able to complete the study, e.g. migrant farm workers,
6. male partner has known erectile or ejaculatory dysfunction,
7. either partner is using any medications or preparation applied topically or intravaginally to the genitalia other than that supplied for the study,
8. either partner is an employee of study sponsor, competitor or affiliated with clinical research center,
9. currently participating in another sexual health clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
The total clinical failure rates for the test and control condoms | 6 weeks
  The total clinical failure rate of a new test condom is comparable with the failure rate of a commercially available latex condom when used during vaginal intercourse as reported by study participant questionnaire.

SECONDARY OUTCOMES:
Clinical / Non-clinical slippage rates acceptability; and Adverse events | 6 weeks
  Evaluate the slippage rates of the polyurethane and the commercially available latex condom when used during vaginal intercourse, as reported by the study participant questionnaire.
Clinical/non-clinical breakage rates | 6 weeks
  Evaluate the breakage rates of the polyurethane and the commercially available latex condom when used during vaginal intercourse, as reported by the study participant questionnaire.
User acceptance | 6 weeks
  Evaluate the user acceptance rates of the polyurethane and the commercially available latex condom when used during vaginal intercourse, as reported by the study participant questionnaire.
Adverse events | 6 weeks
  Evaluate the number of adverse events of the polyurethane and the commercially available latex condom when used during vaginal intercourse, as reported by the study participant questionnaires and study Primary Investigators.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Physicians Research Group, Mesa, Arizona
  - Angels Clinical Research Center, Miami, Florida
  - Physicians Research Group, West Lafayette, Indiana
  - Wellnow, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No